CLINICAL TRIAL: NCT02537002
Title: A Phase 1, Randomized, Double-blind, Sponsor-open, Placebo-controlled, Single Ascending Dose Study To Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of An Intravenous Bolus Infusion Pf-05230907 In Healthy Japanese Subjects
Brief Title: Single Dose Study of PF-05230907 in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B2341003
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: PF-05230907; Pharmacokinetics; Pharmacodynamic; Immunogenicity
MeSH Terms: interventions — PF-05230907

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1- PF-05230907 or Placebo (Experimental)
  Interventions: Drug: PF-05230907; Drug: Placebo
- Cohort 2- PF-05230907 or Placebo (Experimental)
  Interventions: Drug: PF-05230907; Drug: Placebo

INTERVENTIONS:
Drug: PF-05230907 — A single intravenous dose of 3 μg/kg
  Arms: Cohort 1- PF-05230907 or Placebo
Drug: PF-05230907 — A single intravenous dose of 5 μg/kg
  Arms: Cohort 2- PF-05230907 or Placebo
Drug: Placebo — A single intravenous dose of matched placebo

SUMMARY:
The purpose of this study is the following:

* To determine the safety and tolerability of single ascending intravenous (IV) doses of PF-05230907 in healthy Japanese subjects.
* To characterize the PK profile of single ascending IV doses of PF-05230907 in healthy Japanese subjects.
* To characterize the PD profiles of single ascending IV doses of PF-05230907 in healthy Japanese subjects.
* To evaluate the immunogenicity of PF-05230907 in healthy Japanese subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male of females
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs) and <120 kg (265 lbs).
* Japanese subjects who have four biologic Japanese grandparents born in Japan.

Exclusion Criteria:

* Pregnant or nursing females.
* Females of childbearing potential who are unwilling or unable to use an acceptable method of contraception.
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events and Serious Adverse Events Per Participant of PF-05230907 | up to 2 months

SECONDARY OUTCOMES:
Single dose Time to Reach maximum Observed Plasma Concentration (Tmax) of PF-05230907 | Minute 0, 2, 5, 15, 40, 60 minute post-dose
Single dose Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)]of PF-05230907 | Minute 0, 2, 5, 15, 40, 60 minute post-dose
Single dose Plasma Decay Half-Life (t1/2) of PF-05230907 | Minute 0, 2, 5, 15, 40, 60 minute post-dose
Single dose steady state Volume of Distribution (Vss) of PF-05230907 | Minute 0, 2, 5, 15, 40, 60 minute post-dose
Single dose clearance (CL) of PF-05230907 | Minute 0, 2, 5, 15, 40, 60 minute post-dose
Single dose Maximum Observed plasma concentration (Cmax) of PF-05230907 | Minute 0, 2, 5, 15, 40, 60 minute post-dose
Single dose Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (last)]of PF-05230907 | Minute 0, 2, 5, 15, 40, 60 minute post-dose
Change of aPTT from pre-dose to post-dose | Hour 0, 24 hour post-dose
Change of prothrombin fragments 1+2 (PF1+2) | Hour 0, 24 hour post-dose
Change of plasma D-dimer | Hour 0, 48 hour post-dose
Incidence of development of anti-drug antibody (ADA) | up to 2 months
Incidence of development of neutralizing antibody (NAb) | up to 2 months
Change of factor X activity | up to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2341003&StudyName=A%20Phase%201%2C%20Randomized%2C%20Double-blind%2C%20Sponsor-open%2C%20Placebo-controlled%2C%20Single%20Ascending%20Dose%20Study%20To%20Evaluate%20The%20Safety%2C%20Tolerability%2C%20Pharmacokinetics%20And%20Pharmacodynamics%20Of%20An%20Intravenous%20Bolus%20Infusion%20Pf-05230907%20In%20Healthy%20Japanese%20Subjects